CLINICAL TRIAL: NCT04522310
Title: ProAdrenomedullin Assessment of Multi-Organ Failure in COvid-19 Sepsis
Acronym: PAMOCOS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Lens (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-05
Record Dates: First submitted 2020-07-17; First posted 2020-08-21 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — mid-regional pro-adrenomedullin, human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MR-Pro-ADM — Dosage of MR-pro-ADM

SUMMARY:
COVID-19 is a worldwide pandemic. Around 5% of infected patients are admitted in ICU, mainly for respiratory failure. Outcome of these patients is linked to other organ failures. Optimal therapies are not defined so far. The sponsor want to assess the role of MR-ProADM as prognostic biomarker, and the impact of treatments (including supportive treatments) on MOF occurrence and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient admitted in the ICU with COVID-19 pneumonia

Exclusion Criteria:

* Pregnancy
* Legal reasons (patients under guardianship, curatorship)
* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient admitted in the ICU with COVID-19 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Association or correlation between MR-ProADM at day 1 and day 3 and the onset of visceral failures extra respiratory in reanimation. | comparison to day 1 and day 3
  Association or correlation between MR-ProADM at day 1 and day 3 and the onset of visceral failures extra respiratory in reanimation.
mortality at day 28 and day 90. | admission until day 90
  mortality at day 28 and day 90.

SECONDARY OUTCOMES:
Association between MR-ProADM and mortality at day 28. | admission until day 28
  Association between MR-ProADM and mortality at day 28.
Association or correlation between patient factor or treatment, and the onset or aggravation of visceral failures (day 3 and day 10), evolution until day 28. | admission until day 28
  Association or correlation between patient factor or treatment, and the onset or aggravation of visceral failures (day 3 and day 10), evolution until day 28.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Hospital of Arras, Arras
  - Hospital of Boulogne/mer, Boulogne-sur-Mer
  - Hospital of DOUAI, Douai
  - Hospital of Dunkerque, Dunkirk
  - Hospital Dr Schaffner, Lens
  - Hospital of Roubaix, Roubaix
  - Hospital of Tourcoing, Tourcoing
  - Hospitalier of Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No